CLINICAL TRIAL: NCT04434885
Title: Axial Involvement in Psoriatic Arthritis Cohort
Acronym: AXIS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Assessment of Spondyloarthritis International Society (ASAS) (Unknown); Group for Research and Assessment of Psoriasis and Psoriatic Arthritis (Network)
Responsible Party: Principal Investigator, Denis Poddubnyy, Professor of Rheumatology, Charite University, Berlin, Germany
Other Study IDs: AXIS
Record Dates: First submitted 2020-06-15; First posted 2020-06-17 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Psoriatic arthritis: Patients diagnosed with PsA and fulfilling the classification criteria for PsA with symptom duration of up to 10 years and not receiving biological or targeted synthetic disease modifying antirheumatic drugs (b or tsDMARDs).
  Interventions: Other: Clinical and imaging examination of symptoms and signs suggestive of axial involvement

INTERVENTIONS:
Other: Clinical and imaging examination of symptoms and signs suggestive of axial involvement — Clinical and imaging examination including X-rays and magnetic resonance imaging of sacroiliac joints and spine

SUMMARY:
This is a multinational multicenter cross-sectional study in patients with a definite diagnosis of PsA. The population of interest will consist of 400 adult patients diagnosed with PsA and fulfilling the classification criteria for PsA and not receiving biological or targeted synthetic disease modifying antirheumatic drugs (b or tsDMARDs). Participating rheumatologists are encouraged to include consecutive PsA patients not treated with biologic or a targeted synthetic disease-modifying antirheumatic drug because of their potential impact on active inflammatory changes in the axial skeleton, which will be the focus of the current study. Patients will be recruited prospectively in selected study centres and will undergo study-related examinations including imaging of the axial skeleton (X-rays and magnetic resonance imaging). Collected data will serve as a basis for the judgement on the presence or absence of axial involvement by the local investigator and, independently, by the central study committee.

DETAILED DESCRIPTION:
Background. Involvement of the axial skeleton (of sacroiliac joints and / or spine) is one of the frequent manifestations associated with psoriatic skin disease along with involvement of peripheral musculoskeletal structures (peripheral arthritis, enthesitis, dactylitis), which are usually referred to as psoriatic arthritis (PsA). Depending on the definition used, the prevalence of axial disease varies from 25% to 70% of patients with PsA. There is an urgent need for an evidence-based definition and a unified and widely accepted nomenclature for axial involvement in PsA that would allow defining a homogeneous subgroup of patients in the heterogeneous PsA population.

Aim and study objectives. To develop a data-driven definition of axial involvement in PsA based on cross-sectional evaluation of patients with a diagnosis of PsA fulfilling the CASPAR criteria. The study objectives are: to determine the prevalence of axial involvement in a cohort of patients with PsA; to identify the frequency of imaging findings suggestive of inflammatory involvement of axial skeleton in PsA; to identify factors (clinical, lab, imaging) associated with the presence of axial involvement in PsA.

Study design and study population. This is a multinational multicenter cross-sectional study in patients with a definite diagnosis of PsA. The population of interest will consist of 400 adult patients diagnosed with PsA and fulfilling the classification criteria for PsA and not receiving biological or targeted synthetic disease-modifying antirheumatic drugs (b or tsDMARDs). Participating rheumatologists are encouraged to include consecutive PsA patients not treated with biologic or a targeted synthetic disease-modifying antirheumatic drug because of their potential impact on active inflammatory changes in the axial skeleton, which will be the focus of the current study. Patients will be recruited prospectively in selected study centres and will undergo study-related examinations including imaging of the axial skeleton (X-rays and magnetic resonance imaging). Collected data will serve as a basis for the judgement on the presence or absence of axial involvement by the local investigator and, independently, by the central study committee.

Analysis and study outcomes. The prevalence of axial involvement in a cohort of patients with PsA according to the local and central assessment will be calculated in PsA patients presenting with peripheral involvement (the primary analysis population) as well as in the entire group. The prevalence of axial involvement as assessed by the local investigator in PsA patients presenting with peripheral involvement will be the primary outcome of the study. The agreement between local and central judgements will be analyzed. A sub-analysis of a group presenting without peripheral involvement (i.e., pure axial disease) will be performed. The frequency of imaging findings (on MRI and X-rays) suggestive of inflammatory involvement of axial skeleton (sacroiliac joints and spine) in PsA according to the local and central assessment will be calculated. The agreement between local and central judgements will be analyzed. Parameters associated with the presence of axial involvement in PsA will be explored as well. The diagnostic / classification value of each parameter will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years.
* Definite diagnosis of PsA.
* Fulfilment of the CASPAR criteria for PsA.
* Duration of PsA symptoms ≤10 years.
* Written informed consent.

Exclusion Criteria:

* Unable or unwilling to give informed consent or to comply with the protocol.
* Current or past treatment with biologic or a targeted synthetic disease-modifying antirheumatic drug (DMARDs).
* Contraindications for MRI and/or plain X-ray examination of sacroiliac joints and spine.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population of interest will consist of consecutive adult patients diagnosed with PsA and fulfilling the CASPAR (ClASsification criteria for Psoriatic ARthritis) classification criteria for PsA with symptom duration of up to 10 years and not receiving biological or targeted synthetic disease modifying antirheumatic drugs (b or tsDMARDs). Participating rheumatologists are encouraged to include consecutive PsA patients not treated with biologic or a targeted synthetic disease-modifying antirheumatic drug because of their potential impact on active inflammatory changes in the axial skeleton, which will be the focus of the current study.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
The prevalence of axial involvement by local investigator | Baseline
  The frequency of axial involvement (global judgment) as assessed by the local investigator in PsA patients

SECONDARY OUTCOMES:
The frequency of axial involvement by the central committee | Baseline
  The frequency of axial involvement (global judgment) as assessed by the central clinical committee in PsA patients
The frequency of imaging findings suggestive of axial involvement | Baseline
  The frequency of imaging findings (on MRI and X-rays) suggestive of inflammatory involvement of axial skeleton (sacroiliac joints and spine) in PsA according to the local and central assessment

CONTACTS AND LOCATIONS:
Overall Officials: Denis Poddubnyy, MD, Study Chair — Charite University, Berlin, Germany; Dafna D. Gladman, MD, FRCPC, Study Chair — University of Toronto
Locations (2):
- Toronto Western Hospital, Toronto, Ontario, Canada
- Charité - Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Study data will be made available for subsequent analysis upon reasonable request
Supporting Information: Study Protocol
Time Frame: After completion of the primary analysis
Access Criteria: Submission of a research proposal and approval by the study chairs

REFERENCES:
- [Derived] Poddubnyy D, Baraliakos X, Van den Bosch F, Braun J, Coates LC, Chandran V, Diekhoff T, van Gaalen FA, Gensler LS, Goel N, Gottlieb AB, van der Heijde D, Helliwell PS, Hermann KGA, Jadon D, Lambert RG, Maksymowych WP, Mease P, Nash P, Proft F, Protopopov M, Sieper J, Torgutalp M, Gladman DD. Axial Involvement in Psoriatic Arthritis cohort (AXIS): the protocol of a joint project of the Assessment of SpondyloArthritis international Society (ASAS) and the Group for Research and Assessment of Psoriasis and Psoriatic Arthritis (GRAPPA). Ther Adv Musculoskelet Dis. 2021 Dec 18;13:1759720X211057975. doi: 10.1177/1759720X211057975. eCollection 2021. PMID 34987619